CLINICAL TRIAL: NCT05702970
Title: Beneficial Effects of Vitamin D Combined With Oral Iron Supplementation in Patients With Chronic Heart Failure and Iron Deficiency
Acronym: VICTORID-HF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VICTORID-HF
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Iron-deficiency; Heart Failure, Systolic; Heart Failure NYHA Class II; Heart Failure NYHA Class III; Vitamin D Deficiency
Keywords: Heart Failure; Iron Deficiency; Sucrosomial Iron; Ferric Carboxymaltose; Vitamin D
MeSH Terms: conditions — Heart Failure; Anemia, Iron-Deficiency; Heart Failure, Systolic; Vitamin D Deficiency; Iron Deficiencies | interventions — sucrosomial iron; Vitamin D; ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: Interventional, randomized, controlled, open-label, sequential recruitment study
Who Masked: Outcomes Assessor
Masking Description: Patients and examining physicians will be aware of the allocated arm, whereas, outcome analysts will be kept blinded to the treatment allocation arm. This will be accomplished by blinding the investigators assessing: NHYA class, distance walked at 6MWT, KCCQ, vital signs. Echocardiography data will be measured offline or by an independent physician, blinded to the treatment allocation. Events at follow-up will be assessed by an adjudication committee blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ferric Carboxymaltose (Active Comparator): Control Group
  Interventions: Drug: Ferric Carboxymaltose 50 MG/ML
- Sucrosomial iron (Experimental): Experimental arm 1
  Interventions: Drug: Sucrosomial iron
- Sucrosomial iron and vitamin D (Experimental): Experimental arm 2
  Interventions: Drug: Sucrosomial iron; Drug: Vitamin D

INTERVENTIONS:
Drug: Sucrosomial iron — Sucrosomial iron group: administration of sucrosomial iron (SiderAl Forte®) at a dose of 60 mg (2 tablets) once a day for 24 weeks.
  Other Names: SiderAl Forte
  Arms: Sucrosomial iron; Sucrosomial iron and vitamin D
Drug: Vitamin D — administration Vitamin D3 (100,000 IU load at time 0, then 2,000 IU daily) for 24 weeks in combination with of sucrosomial iron (SiderAl Forte®) at a dose of 60 mg (2 tablets) once daily in Sucrosomial iron and vitamin D group
  Other Names: DiBase / UltraD3
  Arms: Sucrosomial iron and vitamin D
Drug: Ferric Carboxymaltose 50 MG/ML — Control group [standard of care]: administration of FCM (Ferinject®) with a dose between 500 and 2000 mg (depending on body weight and Hb values), to be administered in 1 or 2 doses (time 0 ± 6 weeks) with possible additional administration of 500 mg at week 12 in case of persistent ID.
  Other Names: Ferinject
  Arms: Ferric Carboxymaltose

SUMMARY:
The goal of this randomized, controlled, open-label, interventional study is to evaluate whether, in patients with heart failure (HF) and iron deficiency (ID), the administration of vitamin D in combination with sucrosomial iron is as effective as intravenous ferric carboxymaltose in improving symptoms of HF.

The main hypothesis which the study aims to test is the non-inferiority of sucrosomial iron (± vitamin D) compared with FCM treatment, after 24 weeks. Primary endpoint: the performance of the Six-Minute Walking Test, comparing the mean difference from baseline of the distance walked by patients in meters.

Participants will be evaluated in outpatient scheduled visits at 6, 12 and 24 weeks, performing blood tests, clinical evaluation, instrumental investigations and recording any adverse events, cardiovascular events, re-hospitalizations and fractures.

The study will involve randomization into 3 groups with a 1:1:1 ratio:

1. Control group [standard of care]: administration of FCM (Ferinject®) with a dose between 500 and 2000 mg (depending on body weight and hemoglobin values), to be administered in 1 or 2 doses (time 0 ± 6 weeks) with possible additional administration of 500 mg at week 12 in case of persistent ID.
2. Sucrosomial iron group: administration of sucrosomial iron (SiderAl Forte®) at a dose of 60 mg (2 tablets) once a day for 24 weeks.
3. Sucrosomial iron and vitamin D group: administration of sucrosomial iron (SiderAl Forte®) at a dose of 60 mg (2 tablets) once daily + vitamin D3 (100,000 IU load at time 0, then 2,000 IU daily) for 24 weeks

DETAILED DESCRIPTION:
Chronic heart failure (HF) is associated, in more than one third of patients, with iron deficiency (ID), and this comorbidity can have a negative impact on quality of life and survival.

Treatment of ID is recommended in patients with HF and left ventricle ejection fraction (LVEF) <45% to improve symptoms and reduce rehospitalizations.

Intravenous iron supplementation with ferric carboxymaltose (FCM), has been shown to be effective in correcting ID and improving symptoms in patients with HF, therefore, it is considered the standard of care. However, intravenous supplementation is not riskless. The main side effects are as follows:

1. accumulation of circulating non-transferrin bound iron (NTBI), which can lead to increased oxidative stress.
2. increased blood levels of the biologically active form of fibroblast growth factor-23 (FGF-23), especially with the use of FCM. When elevated, this hormone reduces renal phosphate uptake, leading to hypophosphatemia and, consequently, osteomalacia. In patients with chronic kidney disease (CKD), elevated FGF-23 levels have also been associated with left ventricular hypertrophy, myocardial fibrosis, increased adverse cardiovascular events and all-cause mortality, regardless of traditional cardiovascular risk factors.

Oral iron supplementation could therefore be safer in patients with HF, reducing oxidative stress and the risk of altered bone metabolism. To date, the only trial that has evaluated the efficacy of oral iron in HF has provided discouraging data. More precisely, hepcidin inhibition on iron intestinal absorption appears to be the most relevant factor affecting the efficacy of iron treatment.

To overcome hepcidin blockade, it has been proposed to use specific oral iron formulations, which are less susceptible to inhibition of hepcidin (such as sucrosomial iron), and a single high-dose daily administration. Additionally, the possibility of actively reducing hepcidin levels has been explored by administering compounds that act as hepcidin inhibitors. Among these compounds, one of the most promising is vitamin D.

The main hypothesis which the study aims to test is the non-inferiority of sucrosomial iron (± vitamin D) compared with FCM treatment, after 24 weeks. Primary endpoint: the performance of the Six-Minute Walking Test, comparing the mean difference from baseline of the distance walked by patients in meters.

Study design

Interventional, randomized, controlled, open-label, sequential recruitment study of outpatients, diagnosed with symptomatic chronic HF (New York Heart Association - NYHA class II-III), LVEF≤45%, ID (ferritin <100 ng/ml or transferrin saturation - TSAT <20% in case of ferritin levels between 100 and 300 ng/ml) and hemoglobin (Hb) values between 9.5-13.5 g/dL.

In patients hospitalized for acute HF (inpatients), pre-randomization will be performed and re-evaluation for recruitment during outpatient visit will be scheduled at least 3 weeks after discharge.

The study will involve randomization into 3 groups with a 1:1:1 ratio:

1. Control group [standard of care]: administration of FCM (Ferinject®) with a dose between 500 and 2000 mg (depending on body weight and Hb values), to be administered in 1 or 2 doses (time 0 ± 6 weeks) with possible additional administration of 500 mg at week 12 in case of persistent ID.
2. Sucrosomial iron group: administration of sucrosomial iron (SiderAl Forte®) at a dose of 60 mg (2 tablets) once a day for 24 weeks.
3. Sucrosomial iron and vitamin D group: administration of sucrosomial iron (SiderAl Forte®) at a dose of 60 mg (2 tablets) once daily + Vitamin D3 (100,000 IU load at time 0, then 2,000 IU daily) for 24 weeks

Period of treatment and follow-up The expected duration of subject participation is approximately 27 weeks. The duration of the screening period is up to 3 weeks (although may be longer for subjects rescreened); treatment period is 24 weeks.

During treatment, patients will be evaluated in outpatient scheduled visits at 6, 12 and 24 weeks, performing blood tests, clinical evaluation, instrumental investigations and recording any adverse events, cardiovascular events, re-hospitalizations and fractures.

After completion of treatment, an echocardiographic evaluation will also be performed to assess parameters of systolic and diastolic function, parietal thicknesses, and left ventricular diameters.

Hypothesis Formulation and Testing Procedure The three-arm design with two experimental treatments poses the need to evaluate the effects of sucrosomial iron treatments before comparing them with FCM. The investigators decided to base the comparison of sucrosomial iron with FCM on the results of the non-inferiority test between the two experimental treatments (first non-inferiority test; NIT1). Let's SI= sucrosomial Iron; SID=sucrosomial Iron + Vitamin D; FCM: Ferric carboxymaltose; if non-inferiority is assessed, the investigators will test the pooled experimental group (SID+SI) against the FCM group (second non-inferiority test, version A; NIT2-A), otherwise the investigators will interrupt the study. In the case of the superiority of SID over SI, the investigators will test the non-inferiority of SID (not pooled) over the control treatment (second non-inferiority test, version B; NIT2-B). An interim analysis for NIT1 will be performed at the half of patient enrolment to assess whether to stop for efficacy/futility or continue in patients' enrolment

Assumption and sample size The investigators have information from the CONFIRM-HF study that compared the 6MWT-as difference from baseline-of FCM group versus placebo. The FCM group, after 24 weeks, walked an average of 18 meters more than at the baseline, with a standard deviation of 8, while the placebo group walked an average of 16 meters less than at the baseline, with an equal standard deviation of 8. Thus, the investigator assume a standard deviation of 8, equal for the three arms. The ΔNIT1 has been fixed to 3.2 meters and ΔNIT2 equal to 7. Finally, assuming 80% of power, 5% Type I error for both NIT1 and NIT2 (since they have a hierarchical structure), the sample size required for NIT1 is 234. After accounting for potential dropouts (10%), the final calculated sample size is 258 that is adequate to conduct also the subsequent noninferiority hypothesis test, in any case (NIT2-A or NIT2-B)

ELIGIBILITY:
Inclusion Criteria:

NYHA functional class II-III due to symptomatic chronic HF and all the following:

* At least 3 weeks since the last hospitalization or emergency department access for acute HF decompensation.
* Optimal drug treatment for HF according to the European Society of Cardiology guidelines determined by the investigator (unless contraindications or treatment not tolerated).
* No changes in HF therapy dosage in the previous 2 weeks (except diuretics).
* No new HF therapy in the 3 weeks prior to recruitment.
* LVEF ≤45%.
* Brain Natriuretic Peptide (BNP) >100 pg/mL and/or NT-proBNP >400 pg/mL at pre-recruitment evaluation.
* Evidence of ID defined as ferritin <100 ng/ml or TSAT <20% in case of ferritin levels between 100 and 300 ng/ml.
* 25-OH-Vitamin D levels <50 nmol/L.
* The subject must be able to complete the 6MWT.
* At least 18 years of age.

Exclusion Criteria:

* Myocardial infarction or acute coronary syndrome, transient ischemic attack or stroke, coronary artery bypass, percutaneous intervention, or major thoracic or cardiac surgery within the previous 2 months.
* Clinically relevant (severe) non-corrected valvular heart disease, obstructive cardiomyopathy.
* Chronic anemia due to non-correctable causes other than ID and anemia of chronic disease (e.g., hemoglobinopathies, hematologic malignancies, hemolytic anemia).
* Anemia due to Vitamin B12 or acid folic deficiency. Recruitment may be re-evaluated at least 6 weeks after the end of vitamin B12 and or folic acid supplementation.
* History of acquired iron overload.
* Administration of erythropoietin, iron supplementation (either oral or intravenous iron), blood transfusion in the previous 6 weeks or already scheduled for the 3 months after recruitment.
* Administration of vitamin D or similar in the 3 months preceding or already scheduled for the 3 months following recruitment.
* Severe bone disease.
* Active infections, C-reactive protein (CRP) >20 mg/L, clinically significant bleeding, active neoplasm (with exception of basal cell or squamous cell carcinoma of the skin and intraepithelial cervical neoplasia).
* Chronic liver disease (including active hepatitis) and/or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3x normal limit.
* Immunosuppressive therapy or dialysis.
* Pregnancy or breastfeeding.
* The subject has a known sensitivity to any of the products that will be administered during the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of Six-Minute Walking Test (6MWT) | 24 weeks
  To evaluate the change from baseline performance of the 6MWT, in the three treatment arms, measuring the distance walked by patients in meters

SECONDARY OUTCOMES:
Quality of life (QoL) assessment | 24 weeks
  To evaluate the change from baseline in the Kansas City Cardiomyopathy Questionnaire (KCCQ) in the three treatment arms
Cardiovascular and general endpoint 1 | 12 and 24 weeks
  Change from baseline in the NYHA class in the sucrosomial iron + vitamin D group compared with the control group
Cardiovascular and general endpoint 2 | 12 and 24 weeks
  Change from baseline in the NYHA class in the sucrosomial iron + vitamin D group compared the sucrosomial iron group
Cardiovascular and general endpoint 3 | 12 and 24 weeks
  Change from baseline in distance walked at 6MWT in the sucrosomial iron + vitamin D group compared with sucrosomial iron alone
Cardiovascular and general endpoint 4 | 12 and 24 weeks
  Change in the glomerular filtration rate estimated using the CKD-EPI formula.
Cardiovascular and general endpoint 5 | 12 and 24 weeks
  Surviving days out of hospital.
Cardiovascular and general endpoint 6 | 12 and 24 weeks
  Hospitalizations (total, cardiovascular, due to HF).
Cardiovascular and general endpoint 7 | 12 and 24 weeks
  Mortality (total, cardiovascular, due to HF)
Echocardiographic endpoint 1 | 24 weeks
  Changes in left ventricle ejection fraction [LVEF, Simpson's method] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 2 | 24 weeks
  Changes in left ventricle end diastolic diameter [LVEDD] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 3 | 24 weeks
  Changes in left ventricle end systolic diameter [LVESD] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 4 | 24 weeks
  Changes in left ventricle end diastolic volume [LVEDV] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 5 | 24 weeks
  Changes in left ventricle end systolic volume [LVESV] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 6 | 24 weeks
  Changes in Interventricular septal thickness [IVS] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 7 | 24 weeks
  Changes in left ventricular posterior wall [PW] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 8 | 24 weeks
  Changes in diastolic function [E/e'] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 9 | 24 weeks
  Changes in diastolic function [E/A ratio] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 10 | 24 weeks
  Changes in left atrial volume index [LAVI] compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 11 | 24 weeks
  Changes in Tricuspid regurgitation [TR] peak velocity compared with baseline in the sucrosomial iron + vitamin D group
Echocardiographic endpoint 12 | 24 weeks
  Changes in left ventricle ejection fraction [LVEF, Simpson's method] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 13 | 24 weeks
  Changes in left ventricle end diastolic diameter [LVEDD] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 14 | 24 weeks
  Changes in left ventricle end systolic diameter [LVESD] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 15 | 24 weeks
  Changes in left ventricle end diastolic volume [LVEDV] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 16 | 24 weeks
  Changes in left ventricle end systolic volume [LVESV] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 17 | 24 weeks
  Changes in Interventricular septal thickness [IVS] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 18 | 24 weeks
  Changes in left ventricular posterior wall [PW] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 19 | 24 weeks
  Changes in diastolic function parameters [E/A ratio] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 20 | 24 weeks
  Changes in diastolic function parameters [E/e'] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 21 | 24 weeks
  Changes in left atrial volume index [LAVI] in the sucrosomial iron + vitamin D group compared with the control group
Echocardiographic endpoint 22 | 24 weeks
  Changes in Tricuspid regurgitation [TR] peak velocity in the sucrosomial iron + vitamin D group compared with the control group
Calcium-phosphorus metabolism endpoint 1 | 12 and 24 weeks
  Plasma levels of calcium in the sucrosomial iron + vitamin D group compared with the control group
Calcium-phosphorus metabolism endpoint 2 | 12 and 24 weeks
  Plasma levels of phosphate in the sucrosomial iron + vitamin D group compared with the control group
Calcium-phosphorus metabolism endpoint 3 | 12 and 24 weeks
  Plasma levels of FGF-23 in the sucrosomial iron + vitamin D group compared with the control group
Calcium-phosphorus metabolism endpoint 4 | 12 and 24 weeks
  Plasma levels of calciumin the sucrosomial iron group compared with the control group
Calcium-phosphorus metabolism endpoint 5 | 12 and 24 weeks
  Plasma levels of phosphate in the sucrosomial iron group compared with the control group
Calcium-phosphorus metabolism endpoint 6 | 12 and 24 weeks
  Plasma levels of FGF-23 in the sucrosomial iron group compared with the control group
Calcium-phosphorus metabolism endpoint 7 | 12 and 24 weeks
  Incidence of fractures in the sucrosomial iron + vitamin D group compared with the control group
Calcium-phosphorus metabolism endpoint 8 | 12 and 24 weeks
  Incidence of fractures in the sucrosomial iron group compared with the control group

CONTACTS AND LOCATIONS:
Overall Officials: Federico Capone, MD, Principal Investigator — University of Padova; Roberto Vettor, MD, Study Director — University of Padova

IPD SHARING:
Plan to Share IPD: Undecided